CLINICAL TRIAL: NCT06939855
Title: Efficacy and Safety of QL1706 in the Treatment of Advanced Bone and Soft Tissue Sarcoma: a Phase II Clinical Study
Brief Title: QL1706 in the Treatment of Advanced Bone and Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Wang,MD, Department of Bone and soft tissue Oncology, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-200-X01
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bone and Soft Tissue Tumors
Keywords: QL1706
MeSH Terms: conditions — Soft Tissue Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental：QL1706 (Experimental): Drug QL1706
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4)

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — 5mg/kg iv q3w

SUMMARY:
This is a single-center, open-label phase II study of QL1706 for the treatment of advanced bone and soft tissue sarcomas.The study includes screening period, treatment period and follow-up period. Subjects will receive QL1706 5mg/kg iv every 3 weeks until disease progression or intolerance. Efficacy should be evaluated and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the study, sign the informed consent form (ICF), and are able to comply with study procedures.
2. Age ≥18 years and ≤75 years at the time of signing ICF, regardless of gender.
3. Histologically confirmed unresectable locally advanced or metastatic bone and soft tissue sarcoma at this institution, including: undifferentiated sarcoma, leiomyosarcoma, myxofibrosarcoma, alveolar soft part sarcoma, pleomorphic undifferentiated sarcoma, chordoma, angiosarcoma, and dedifferentiated liposarcoma.
4. For histological subtypes without standard systemic therapy, such as chordoma, prior systemic therapy is not required. Subjects with alveolar soft part sarcoma may be systemic therapy-naïve or have received systemic therapy excluding PD-1/PD-L1 inhibitors.
5. For histological subtypes with standard systemic therapy, such as undifferentiated sarcoma, leiomyosarcoma, myxofibrosarcoma, dedifferentiated liposarcoma, and pleomorphic undifferentiated sarcoma, subjects must have received anthracycline-based chemotherapy. Subjects with angiosarcoma must have received paclitaxel- or anthracycline-based chemotherapy, and have developed metastasis or disease progression (≥10% increase in the sum of the longest diameters within 3 months), or be intolerant to standard therapy.
6. At least one measurable lesion as assessed by the investigator according to RECIST v1.1.
7. Subjects are able to provide tumor tissue samples and blood samples for biomarker testing including PD-L1.
8. ECOG performance status of 0-1, with an expected survival ≥12 weeks.
9. Clinical laboratory tests at screening must meet the following criteria (no use of blood components, hematopoietic growth factors, leukocyte- or platelet-stimulating agents, or anemia-correcting medications within 14 days before testing):

   1. Hematologic: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L; Platelet count (PLT) ≥90 × 10⁹/L; Hemoglobin (Hb) ≥90 g/L.
   2. Hepatic function: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN); for subjects with liver metastasis, AST and ALT ≤5 × ULN. Total bilirubin (TBIL) ≤1.5 × ULN (subjects with Gilbert syndrome: TBIL <3 × ULN). Albumin (ALB) ≥30 g/L.
   3. Renal function: Serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance (CCr) ≥50 mL/min (calculated by Cockcroft-Gault formula).
   4. Coagulation: Activated partial thromboplastin time (APTT) ≤1.5 × ULN; International normalized ratio (INR) ≤1.5; Prothrombin time (PT) ≤1.5 × ULN.
   5. Urine protein: Urine protein dipstick ≤1+. If ≥2+, a 24-hour urine protein test is required; subjects with <1 g/day are eligible.
   6. Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%.
10. Female subjects must be non-lactating, and a pregnancy test must be negative before enrollment.
11. Subjects of childbearing potential agree to use effective contraception from signing the ICF through at least 180 days after the last dose of study drug.

Exclusion Criteria:

1. Known history of severe allergic reactions to any monoclonal antibody or any excipient in its formulation.
2. Currently participating in and receiving investigational treatment, or participation in an investigational drug/device study with investigational treatment administered within 4 weeks before the first dose of study treatment.
3. History of other active malignancies within 5 years prior to first dose. Cured localized malignancies such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, cervix, or breast are not restricted by time.
4. Prior treatment with immune checkpoint inhibitors (PD-1/PD-L1 agents) or other agents targeting T-cell receptor signaling (for example CTLA-4, OX-40). Subjects treated more than 5 years earlier and with no clinical evidence of disease recurrence within the past 5 years may be eligible.
5. Presence of brain metastasis. Subjects with asymptomatic brain metastasis or symptomatic metastasis that is stable for ≥4 weeks after treatment may be enrolled.
6. Active autoimmune disease requiring systemic therapy (disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to enrollment. Conditions include but are not limited to myasthenia gravis, systemic lupus erythematosus, interstitial lung disease, uveitis, ulcerative colitis, autoimmune hepatitis, hypophysitis, systemic vasculitis, nephritis, hyperthyroidism, hypothyroidism, mixed connective tissue disease. Subjects with vitiligo or fully resolved childhood asthma without intervention in adulthood are eligible. Asthma requiring bronchodilator therapy is not eligible. Physiologic replacement therapy (thyroxine, insulin, or corticosteroids for adrenal or pituitary insufficiency) is not considered systemic therapy.
7. Active pulmonary tuberculosis, radiation pneumonitis, drug-induced pneumonitis, or other significant pulmonary impairment during screening.
8. Requirement for long-term or high-dose nonsteroidal anti-inflammatory drugs (aspirin ≥325 mg) or anticoagulant therapy.
9. Clinically significant gastrointestinal disorders including, but not limited to, history of gastrointestinal bleeding or perforation, or acute pancreatitis.
10. Cardiovascular or cerebrovascular diseases including:

(1) Heart failure ≥NYHA class II. (2) Severe or unstable angina. (3) Myocardial infarction or cerebrovascular accident within 6 months before first dose, or aortic aneurysm requiring surgical repair.

(4) Atrial fibrillation or clinically significant supraventricular/ventricular arrhythmias requiring treatment.

(5) Symptomatic superior vena cava syndrome. (6) QTc >450 ms (male) or QTc >470 ms (female). (7) Hypertension not adequately controlled with medication (systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg), or history of hypertensive crisis or hypertensive encephalopathy.

11. Hereditary or acquired bleeding tendency or coagulation disorders. 12. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage.

13. Active infection or unexplained fever >38.5°C during screening. Fever confirmed to be cancer-related may be eligible.

14. Use of broad-spectrum antibiotics by any route within 30 days before first dose.

15. Systemic corticosteroid therapy (≥10 mg/day prednisone or equivalent) or other immunosuppressants (such as cyclosporine, cyclophosphamide, azathioprine, methotrexate, thalidomide) within 14 days before first dose, or use of immunostimulatory agents (such as interferons or interleukin-2) within 4 weeks.

16. Major surgery without fully recovered wound healing, severe fractures, therapeutic clinical trial, or traditional Chinese medicine treatment within 4 weeks before first dose; or use of traditional Chinese medicine within 2 weeks.

17. Adverse events from prior antitumor therapy not recovered to ≤Grade 1 (alopecia and cancer-related fatigue excepted, neurotoxicity allowed ≤Grade 2).

18. HIV infection, other acquired or congenital immunodeficiencies, or history of organ or allogeneic bone marrow transplantation (corneal transplantation excepted).

19. Positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis B core antibody (HBcAb) with HBV DNA >1×10⁴ copies/mL (approximately >2000 IU/mL); or positive hepatitis C antibody (HCV-Ab) with HCV-RNA >1×10³ copies/mL. Subjects with dual positivity for HBsAg and HCV-RNA are excluded.

20. Receipt of live or attenuated vaccines within 30 days prior to first dose. 21. Known psychiatric disorders, epilepsy, dementia, or alcohol/drug abuse that may affect compliance.

22. Any condition including medical history, concomitant disease, treatment, or abnormal laboratory results that may confound study results, interfere with participation, or deemed not in the best interest of the subject by the investigator or sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
12 week PFS | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs earlier, assessed at 12 weeks after first treatment
  The PFS rate at 12 weeks after the first injection assessed by the the investigator according to RECIST V1.1

SECONDARY OUTCOMES:
overall response rate (ORR) | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 2 years
  The ORR assessed by the investigator according to RECIST V1.1
The Disease Control Rate (DOR) | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 2 years
  The DOR assessed by the investigator according to RECIST V1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No